CLINICAL TRIAL: NCT04244279
Title: The Efficacy of Ergonomic Intervention in Preventing Musculoskeletal Disorders Among Women After Giving Birth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Prof. Mordechai Dulitzky, Head of obstetrics at Sheba Medical Center, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SHEBA-19-6259-MD-CTIL
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Musculoskeletal Disorders; Musculoskeletal Pain; Post Partum
Keywords: De Quervain syndrome; Low back pain; Neck pain; Wrist pain
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain; Low Back Pain; Neck Pain | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: A comparative experimental study will be conducted with a sample of 50 postnatal women, divided into two groups: 1. An intervention group that will be sampled in a convenience sample. 2. A control group that will be matched to the intervention group according to maternal age and number of children.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All the he REBA assessment will be analyzed by a therapist who is blinded to the participants group belonging.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will participate in a workshop regarding ergonomic principles in baby care. Finally, a brochure will be distributed summarizing the main contents of the workshop. One month and two months after the intervention, the intervention group will receive a videotaped reminder of the principles presented at the workshop via an email or WhatsApp message.
  Interventions: Other: Ergonomic workshop; Other: Brochure; Other: Videos
- Control group (No Intervention): The control group will not receive any intervention during the data collection period. The intervention will be given three months after the beginning of the research, in the format of the brochure and videos sent via email or WhatsApp.

INTERVENTIONS:
Other: Ergonomic workshop — Participants will participate in a single meeting workshop regarding ergonomic principles in baby care.
  Arms: Intervention group
Other: Brochure — Participant will receive a brochure summarizing the main contents of the workshop.
  Arms: Intervention group
Other: Videos — During the next three months after the beginning of the research, they will receive videos that will be a reminder of the principles learned in the workshop.
  Arms: Intervention group

SUMMARY:
The woman's body undergoes many physiological changes during pregnancy, which can cause muscle weakness and postpartum joint instability. In addition, the intensive care of the baby sometimes involves extreme body postures and mechanical loading on the hands, which are considered as ergonomic risk factors. Therefore, postpartum women may be particularly vulnerable to musculoskeletal disorders (MSDs). As far as we know, there is no evidence-based intervention on this issue.

DETAILED DESCRIPTION:
The study will be conducted in the Obstetrics Departments at the Sheba Medical Center. After approval by the Helsinki Committee at the Medical Center all subjects who meet the inclusion criteria will be asked to sign an informed consent form for participation in the study.

The first data collection point will be in the early days after birth, when the subjects are still hospitalized. All the subjects will fill out a demographic questionnaire and two more questionnaires regarding the prevalence and intensity of MSD. The REBA, a standardized observation will be conducted to identify the level of ergonomic risk during the performance of two tasks of baby care .

The REBA will be analyzed by a therapist who is blinded to the participants group belonging.

The participants will be assigned into two groups, intervention group and control group. Number of birth and participant age will be adjusted between the groups. The intervention group will participate in a workshop regarding ergonomic principles in baby care. A brochure will be distributed summarizing the main contents of the workshop. One month and two months after the intervention, participants in the intervention group will receive a videotaped reminder of the principles presented at the workshop via an email or WhatsApp message, along with a request to report the intensity of pain. The control group will not receive the intervention at this time but will also be asked to fill in the scale at the same time points.

Three months after delivery, all subjects will complete the questionnaires regarding the prevalence and intensity of MSD. The REBA will be performed in order to identify the ergonomic risk level during the performance of the same two tasks of baby care. At this point, the control group will receive the intervention in the format of the brochure and videos sent via email or WhatsApp.

The final data collection will be six to twelve months after delivery when all subjects will complete the same questionnaires and a recurrent REBA standardized observation in order to identify the ergonomic risk level during the performance of the same two baby-care tasks will be performed for the last time.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-40
* Hospitalized in a maternity ward in a hospital after the birth of one baby
* Delivery occurred after 37 weeks' gestation

Exclusion Criteria:

* Women with previous orthopedic or rheumatic problems
* Women with neuropathic problems due to non-gestational diabetes
* Women with neurological diseases.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the level of risk factors that result from poor body postures when carrying and feeding the baby. | We will measure three outcomes: Pre-intervention scores (Base-line): During the first meeting in the hospital, after signing a consent form. Follow up 1 and 2:Three months and Six to twelve months after the first meeting.
  This outcome measure will be determined by the Rapid Entire Body Assessment (REBA). A posture analyze assessment for evaluating workloads that are at risk for developing musculoskeletal problems. This measure divides the body into 6 areas that are individually encoded and relates to changes in muscle activity that occur due to static, dynamic, unstable, or variable posture (Al Madani & Dababneh, 2016). The final risk score ranges from 1 (minimum) to 15 (maximum) (Ratzon and Schechter-Margalit, 2007), and the final score describes 5 levels of risk that relate to the need for intervention, with 1 meaning "no need for intervention" and 5 means "immediate need for intervention. "(Al Madani & Dababneh, 2016). This assessment tool is commonly used in the field of ergonomics.
The change in the prevalence of musculoskeletal pain | We will measure three outcomes: Pre-intervention scores (Base-line): During the first meeting in the hospital, after signing a consent form. Follow up 1 and 2:Three months and Six to twelve months after the first meeting.
  This outcome measure will be determined by the Standardized Nordic questionnaire for the analysis of musculoskeletal symptoms (SNQ). The tool is designed for self-filling or for use as an interview (Kuorinka et al., 1987). It is divided into 9 anatomical areas that include the neck, shoulders, elbow, wrist, upper back, lower back, hip, knee and ankle. For each area, there are 3 yes / no questions that relate to the presence of musculoskeletal pain in the last 12 months and 7 days, and to having a functional limitation due to their presence in each area.Ratzon & Mizrachi (2008), added an extension to a questionnaire that included the arm, forearm, palm, and each finger. This supplement was found as valid against the Disabilities of the Arm Shoulder and Hand Questionnaire (DASH) which is moderately correlated with the original SNQ questionnaire (Ratzon & Mizrachi, 2008).
The change in the intensity of musculoskeletal pain | We will measure five outcomes: Pre-intervention(Base-line): During the first meeting in the hospital, after signing a consent form. Follow up 1,2,3 and 4: One month, Two months, Three months and Six to Twelve months after the first meeting.
  This outcome measure will be determined by the Numeric rating scale (NRS). A tool for measuring the intensity of pain in adults. It is a numerical version of The Visual Analog Scale (VAS). The subject is asked to select a number from 0 to 10 which best reflects the current pain intensity he has felt in the last 24 hours, relative to 13 different anatomical regions. The scale is shown in the horizontal line with the number 0 meaning "not painful" and the number 10 meaning "very painful".

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided